CLINICAL TRIAL: NCT03742921
Title: ISTODAX® for Intravenous Infusion 10mg Drug Use Results Survey - Relapsed or Refractory Peripheral T-Cell Lymphoma
Brief Title: ISTODAX® for Intravenous Infusion Drug Use Results Survey- Relapsed or Refractory Peripheral T-Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: ROMI-PTCL-001; U1111-1222-2854 (Registry Identifier: WHO)
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Lymphoma, T-Cell, Peripheral
Keywords: Istodax; Survey; Relapsed or refractory; Peripheral T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Recurrence | interventions — romidepsin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Relapsed or Refractory T-Cell Lymphoma patients with Istodax: Among patients with relapsed or refractory peripheral T-Cell lymphoma, patients who received Istodax will be targeted in this surveillance
  Interventions: Drug: Istodax

INTERVENTIONS:
Drug: Istodax — Istodax

SUMMARY:
To ascertain the safety and efficacy of Istodax® in actual clinical settings in patients with relapsed or refractory peripheral T-cell lymphoma (PTCL) who receive Istodax.

1. Planned registration period 4 years
2. Planned surveillance period 5 years and 6 months

ELIGIBILITY:
Inclusion Criteria:

- Patients who have been diagnosed with relapsed or refractory PTCL who receive Istodax for the first time.

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Since the number of patients with PTCL was 48 and 131 in the Japanese and overseas clinical studies, respectively, the number of subjects to be surveyed was established at 130 to allow comparison of results between this survey and Japanese clinical study, or between this survey and overseas clinical study.
  Among events that were established as the key survey items of this survey, QT interval prolonged had the lowest incidence (3.8%) in the overseas/Japanese clinical studies of Istodax in patients with PTCL. When 130 subjects are collected, it would be possible to collect at least 1 case of an event that occurs at the frequency of 2.3% with a reliability of 95%. Thus, assuming that adverse events occur under the actual use conditions at similar frequencies as in clinical studies, it would be possible to obtain at least 1 case of all events that have been established as the key survey items.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to approximately 5 years
  Number of participants with adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Jinshu Cho, MD, Study Director — Celgene
Locations (1):
- Nihon Seimei Hospital, Osaka, Japan